CLINICAL TRIAL: NCT02816957
Title: Study of The Therapeutic Benefits of Nigella Sativa in Children With Beta Thalassemia Major
Brief Title: Benefits of Nigella Sativa in Children With Beta Thalassemia Major
Acronym: Nigella
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30794l03l16
Record Dates: First submitted 2016-06-23; First posted 2016-06-29 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2016-06

CONDITIONS: Nigella Sativa With Beta Thalassemia Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients receiving Nigella (Active Comparator): 40 patients in the treatment group that will receive nigella sativa powder (2 gm/day) for 3 consecutive months.
  Interventions: Drug: nigella sativ
- patients not received nigella as controls (No Intervention): 40 patients in the control group will not receive nigella sativa and continued on the usual chelators

INTERVENTIONS:
Drug: nigella sativ — nigella sativa powder (2 gm/day) for 3 consecutive months.
  Arms: patients receiving Nigella

SUMMARY:
Evaluate the therapeutic effects health benefits, and immunological effect of Nigella sativa in children with beta thalassemia major.

DETAILED DESCRIPTION:
Study will be carried on children patients with β- thalassemia major attending The Hematology Unit of Pediatric Department at Tanta University Hospital. patients are divided into 2 groups: patients in the control group, patients in the treatment group that will receive nigella sativa powder for 3 consecutive months. Then Evaluate the therapeutic effects health benefits, and immunological effect of Nigella sativa in children with beta thalassemia major.

Evaluate the extent of clinical improvement, reductions in serum iron and ferritin, antioxidant status, treatment of the causes of hemolysis and other therapeutic benefits of Nigella sativa in those patient.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia with iron overload

Exclusion Criteria:

* Thalassemia complicated with diabetes mellitus or hepatitis
* Patients who discontinue treatment

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
malondialdehyde | 3 months
  nmol serum level of malondialdehyde (nmol per liter)
cluster of differentation4 and 8(CD4 and CD8) | 3 months
  CD4 and CD8 cell per cmm
total antioxidant | 3 months
  total antioxidant(mmol per liter)

SECONDARY OUTCOMES:
Serum iron | 3 months
  microgram per dl
total iron binding capacity | 3 months
  microgram per dl
serum ferritin | 3 months
  ng per ml
complete blood count | 3 months
  complete blood count

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ramadan ELshanshory, prof, Study Director — professor of pediatrics
Locations (1):
- Faculty of Medicine- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided